CLINICAL TRIAL: NCT01154062
Title: An Open-label Pilot Study to Evaluate the Safety, Tolerability,Pharmacokinetics, Exploratory Efficacy and Pharmacodynamics of Oral Pazopanib Administered for 28 Days to Neovascular Age-relatedmacular Degeneration Patients
Brief Title: A Study to Evaluate Pazopanib Tablets in Patients Who Have Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114155
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Macular Degeneration
Keywords: age-related macular degeneration; pazopanib; choroidal neovascularization; GW786034
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- low dose (Experimental): Pazopanib tablet
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib tablet

SUMMARY:
A study to evaluate pazopanib tablets in male and female adults of non-child bearing potential with subfoveal CNV due to neovascular AMD. The goal is to assess safety and how well the subjects tolerate the drug. The study will also look at how the body breaks down and metabolizes the drug. All subjects will start the study up to 8 days prior to receiving drug. Once started subjects will take one tablet each day for 28 days. A follow up visit will occur approximately 2 weeks after drug is stopped.

DETAILED DESCRIPTION:
This is a multi-center, open label study of pazopanib administered for 28 days in adult patients with subfoveal CNV due to neovascular AMD. The primary aim is to evaluate safety and tolerability in patients with neovascular AMD and a secondary aim is to evaluate pharmacokinetics and pharmacodynamics. This study does not include a control treatment group (e.g. placebo or active comparator), and instead will be benchmarked to visual acuity and OCT changes observed following treatment with other anti-angiogenic agents in a similar patient population over the same treatment period.

All subjects will receive tablets administered once daily. Subjects will be screened within eight days prior to treatment assignment and initiation of study treatment. The duration of treatment will be 28 days, and subjects will participate in a baseline and four subsequent weekly study visits during the treatment phase. Subjects will also return for a follow-up visit approximately two weeks after last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Age-related macular degeneration patients diagnosed with subfoveal choroidal neovascularization in the study eye, with all of the following characteristics required and confirmed by a central reading center:

  * CNV caused by AMD that extends under the geometric center of the foveal avascular zone
  * CNV comprises ≥ 50% of lesion area
  * Total lesion area no greater than 12 disc areas on fluorescein angiography, where the lesion complex includes CNV, blood, blocked fluorescence not from blood, and serous detachment of the retinal pigment epithelium
  * classic CNV comprises <50% of the lesion area
  * fibrosis comprises ≤ 25% of lesion area
  * Center subfield > 320 microns on SD-OCT (inclusive of subretinal fluid)
  * if no evidence of classic CNV, then presumed to have recent disease progression because of deterioration (≥ 5 letter decrease in vision or evidence of growth of a CNV lesion on fluorescein angiography ) within last 3 months or evidence of hemorrhage from CNV
* Best-corrected ETDRS visual acuity score in the study eye of between 25 and 73 letters (approximately equivalent to Snellen VA of 20/320 to 20/32) at screening.
* Male or female ≥ 50 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential defined as either pre-menopausal with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases of postmenopausal status a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) or value consistent with local laboratory recommended value is confirmatory.
* Subject is willing and able to return for all study visits, and is willing and able to comply with all protocol requirements and procedures.
* Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. If the subject is unable to read the consent form due to visual impairment then the consent must be read to the subject verbatim by person administering the consent, a family member or legally acceptable representative. (Note: Consent by legally acceptable representative is allowed where this is in accordance with local laws, regulations and ethics committee policy.)
* QTcF <450msec; or QTcF<480msec in subjects with Bundle Branch Block.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Additional eye disease in the study eye that could compromise best-corrected visual acuity (e.g. glaucoma with documented visual field loss, clinically significant diabetic retinopathy, ischemic optic neuropathy, infection or retinitis pigmentosa).
* CNV in the study eye due to other causes unrelated to age-related macular degeneration.
* The presence of retinal angiomatous proliferation (RAP) in the study eye, as determined by the investigator (confirmation by indocyanine green angiography is not required).
* Geographic atrophy involving the center of the fovea in the study eye.
* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation of the fundus for photographs, fluorescein angiography and SD-OCT.
* Vitreous, subretinal or retinal hemorrhage in the study eye that is unrelated to AMD. Any previous treatment in the study eye for neovascular AMD, approved or investigational.
* Current intravitreal anti-VEGF therapy in the fellow eye.
* Within 6 months prior to the Screening Visit, use of any systemically administered anti-angiogenic agent (e.g., bevacizumab, sunitinib, cetuximab, sorafenib, pazopanib), approved or investigational.
* Intraocular surgery in the study eye within 3 months of dosing.
* Aphakia or total absence of the posterior capsule (Yttrium aluminum garnet (YAG) capsulotomy permitted) in the study eye.
* History of vitrectomy in the study eye.
* Presence of RPE tear in the study eye.
* Subject has uncontrolled glaucoma (intraocular pressure >25 mmHg) despite treatment with anti-glaucoma medication.
* Within 6 months prior to the Screening Visit, use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol).
* Use of systemic steroids (>10 mg prednisone or equivalent/day) within 14 days of first dose.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).

Medical history or unresolved medical condition, for example:

* Uncontrolled Diabetes Mellitus, with hemoglobin A1c (HbA1c) > 10%
* Myocardial infarction or stroke within 6 months of screening
* Active bleeding disorder
* Major surgery within 3 months of screening
* Hepatic impairment
* Clinically relevant thyroid disease

  * Uncontrolled hypertension, based on criteria provided in Section 4.4.1.2.
  * Subject has a history within the past 2 years of alcohol, substance abuse, or psychiatric disorder likely to confound the efficacy or safety assessments. A history of known HIV infection.
  * Use of prohibited medications listed in Section 9.2 within the restricted timeframe relative to the first dose of study medication.
  * History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
  * A condition or situation, which, in the opinion of the investigator, may result in significant risk to the patient, confound the study results or interfere significantly with participation.
  * History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08-16 (Actual); Primary Completion 2011-04-29 (Actual); Study Completion 2011-04-29 (Actual)

PRIMARY OUTCOMES:
Safety endpoints include complete ophthalmic examination, visual acuity, vital signs (heart rate and blood pressure), clinical laboratory tests, clinical monitoring and adverse event reporting | 1 month

SECONDARY OUTCOMES:
Changes in visual acuity, central retinal thickness, central retinal lesion thickness, retinal morphology, neovascular size, lesion size, and characteristics by fluoresceinangiography and fundus photography. Also, (CL/F), (V/F), (Ka), and (Cτ) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Austin, Texas

REFERENCES:
- [Derived] McLaughlin MM, Paglione MG, Slakter J, Tolentino M, Ye L, Xu CF, Suttle AB, Kim RY. Initial exploration of oral pazopanib in healthy participants and patients with age-related macular degeneration. JAMA Ophthalmol. 2013 Dec;131(12):1595-601. doi: 10.1001/jamaophthalmol.2013.5002. PMID 24113783
- See also: Results for study 114155 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114155?search=study&search_terms=114155#rs